# Georgia State University Informed Consent

**Title:** Passion Daily (Information Session and Daily Surveys)

Principal Investigator: Dominic Parrott, Ph.D.

Sponsor: National Institutes of Health

#### **Introduction and Key Information**

You are invited to take part in a research study. It is up to you to decide if you would like to take part in the study. The purpose of the study is to examine how daily life, including the use of alcohol, affects couples interaction in LGBTQ+ couples. Your role in the study will last over 98 days. On 56 of those days, you will be asked to complete a 5 minute survey. On 42 of those days, you will not be asked to complete the survey. Today's session is an informational session to prepare you for completing the surveys. After today, you will complete a 5 minute survey on requested days using your smart phone. The survey will ask you questions about your social thoughts, behaviors, and past experiences. The risks of being in this study include feeling distress when asked to answer some of these questions. This study is not designed to benefit you. Overall, we hope to gain information about how daily life affects alcohol use and other social thoughts and behaviors in LGBTQ+ couples.

#### **Purpose**

The purpose of the study is to examine how daily life, including the use of alcohol, affects couples interaction in LGBTQ couples. You are invited to take part in this research study because: (1) You endorse a sexual (e.g., bisexual, gay, lesbian, queer) or gender (e.g., trans, non-binary, genderqueer) minority identity, 2) and are in an intimate relationship with a partner, (3) you drink alcohol, (4) you are aged 21 or older, and (5) you are in good health. A total of 900 people will be in this study.

#### **Procedures**

Today's session should last about 45 minutes. If you decide to take part, you and your partner will be seated at a desk. A lab staff member will explain the details of the daily surveys. They will also help you download software on your phone. As part of this research study, you will need to use the LifeData app. When downloading the app, you will be asked to agree to the Terms of Use, which will appear on your mobile device's screen when you begin using the app. If you do not agree to the Terms of Service, you should not take part in this research study. After downloading the app, you will then complete a practice survey. The lab staff member will assist you with this. Starting tomorrow, you will get a "push" notification on your phone each day that reminds you to complete the daily survey. This will occur between 8 a.m. and 12 p.m. for the next 14 days. Then you will have 14 days where you do not need to compete surveys. This process of 14 days of surveys followed by 14 days of no surveys will repeat so that you will have four cycles of surveys (56 days total). Each survey will take no more than 5 minutes to complete. Some of the questions will ask about your partner's behaviors, including questions about behaviors people use when in conflict with their partner. Because both you and your partner must both participate together, this means that your partner will also be asked some questions about your behavior when you both have a conflict with one another. During some of the 14 day breaks

when you are not completing surveys, you may receive messages that provide support and advice for how to deal with stress. Messages will be sent twice a day: one message at 8 a.m. the other at 4 p.m. For each, you will have 4 hours to read it (i.e., until 12 p.m. and 8 p.m.).

## **Future Research**

Researchers will not use or distribute your data for future research studies even if identifiers are removed.

## **Risks**

There is the possibility that participation in this study may cause you some distress when asked to answer certain questions. If you experience distress, you may drop out of the study at any time. There is also a risk that there could be a breach of confidentiality. More information about how we protect your confidentiality is in the confidentiality section below. At the end of the session, we will answer any questions that you may have.

## **Benefits**

If you are randomly assigned to one of the conditions where you receive messages, you may feel supported and learn new ways to deal with stress that are based on empirically supported treatments; however, because this intervention is experimental, we cannot guarantee any benefits. You will receive educational information about alcohol use and couples health. Referrals for alcohol use treatment and mental health counseling will be provided upon request. This information and experience may be seen as benefits. Overall, we hope to gain information about alcohol and other social thoughts and behaviors in LGBTQ+ couples.

#### **Alternatives**

The alternative is to taking part in this study is to not take part in the study.

#### **Compensation**

You will receive \$25 for participating in the study today. You will be paid \$1 for each daily report (up to \$56) plus a bonus based on percent of days complete:

```
52-56 days = $84,
45-51 days (80% complete) = $74,
38-44 days (67% complete) = $64, and
27-37 days (50%) = $54.
```

30 days into the study if you have completed 80% of days, you will receive a \$5 in the form of an e-gift card or cash.

The total possible diary incentives equal \$145 (\$56 + \$84 + \$5). You will be paid every two weeks in the form of an e-gift card or cash.

### **Voluntary Participation and Withdrawal**

You do not have to be in this study. If you decide to be in the study and change your mind, you have the right to drop out at any time. You may skip questions or stop participating at any time. You may refuse to take part in the study or stop at any time, this will not cause you to lose any benefits to which you are otherwise entitled.

## **Confidentiality**

We will keep your records private to the extent allowed by law. The following people and entities will have access to the information you provide:

- Dr. Parrott and his research team
- GSU Institutional Review Board
- Office for Human Research Protection (OHRP)
- National Institutes of Health

We will use a unique number rather than your name on study records. Your data will be stored in locked cabinets and on secure computers. To protect your privacy, the database that links your name and this unique number will be stored separately from these data. Your name will be destroyed in this database within one week of you ending the study. When we present or publish the results of this study, we will not use your name or other data that may identify you. A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time. Questions you answer on the computer will be sent over the internet. Please be aware that data sent over the internet is never entirely secure, but we will take measures to ensure your information is kept safe.

## **Contact Information**

Contact Dominic Parrott at 404-413-6287 or parrott@gsu.edu:

- If you have questions about the study or your part in it
- If you have questions, concerns, or complaints about the study
- If you think you have been harmed by the study

Contact the GSU Office of Human Research Protections at 404-413-3500 or irb@gsu.edu

- if you have questions about your rights as a research participant
- if you have questions, concerns, or complaints about the research

## **Georgia State University Disclaimer**

If you have any question about this study, or believe you have suffered any injury because of participation in the study, you may contact Dr. Dominic Parrott at 404-413-6287. If you have a personal physician, you can request that he/she make available or arrange for appropriate management and treatment for any physical or psychological injury resulting from this study. In the absence of a personal physician, the PI can provide referrals. Georgia State University, however, has not set aside funds to pay for this care or to compensate you if something should

occur. In the unlikely event that you do experience continuing physical or emotional discomfort as a result of this experiment, counseling centers are available to you, including:

Georgia State University Psychology Clinic: 404-413-6229 [sliding fee scale]

Georgia Crisis and Access Line:

1-800-715-4225

Consent

We will give you a copy of this consent form to keep.

If you are willing to volunteer for this research, please sign below.

Printed Name of Participant

Signature of Participant

Date

Principal Investigator or Researcher Obtaining Consent

Date